CLINICAL TRIAL: NCT06740149
Title: Efficacy and Safety of Allogeneic Human Bone Marrow Mesenchymal Stem Cells for the Treatment of Patients with Acute-on-chronic Liver Failure
Brief Title: Efficacy and Safety of BMSCs (CG-BM1) for ACLF Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Cellgenes Biotechnology Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Lin Bingliang, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGBM1-ACLF
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: bone marrow mesenchymal stem cells; acute-on-chronic liver failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 2: Placebo Control (Placebo Comparator): The control group received placebo + conventional treatment. Placebo was solubilizer of CG-BM1. Conventional treatment included hepatoprotection, antiviral therapy or other etiologic treatments, supplementation of plasma and albumin, supplementation of coagulation factors, treatment of complications, and nutritional support.
  Interventions: Drug: Solvent of CG-BM1
- Phase 2: Low Dose Group (Experimental): Patients in low dose group receive CG-BM1 + conventional treatment. Administration procedure of CG-BM1 is 1.0×10^6 cells/kg CG-BM1 once a week for a total of 4 administrations.
  Interventions: Drug: Bone marrow mesenchymal stem cells (low dose)
- Phase 2: Medium Dose Group (Experimental): Patients in medium dose group receive CG-BM1 + conventional treatment. Administration procedure of CG-BM1 is 2.0×10^6 cells/kg CG-BM1 once a week for a total of 4 administrations.
  Interventions: Drug: Bone marrow mesenchymal stem cells (medium dose)
- Phase 1: Low Dose Group (Experimental): The trial group with a low dose (1.0×10^6 cells/kg) will first enroll one subject, who will be infused with single dose CG-BM1 and then observed for at least 28 days. The clinical data of the first subject will be reviewed by the SRC.
  * If the first subject in the low-dose trial group experiences DLT, enrollment will be suspended. After discussion, recommendations will be made. If the trial is to continue, two additional subjects will be enrolled for observation. If no DLT occurs, the dose trial group will need to enroll three more subjects.
  * If the first subject in the dose trial group does not experience DLT after 28 days, - the remaining two subjects in that dose trial group will be enrolled.
  Once all subjects in the dose trial group have completed the infusion and have been observed for 28 days, the clinical data of all subjects will be submitted to the SRC. After a comprehensive evaluation, the SRC will provide recommendations for dose escalation.
  Interventions: Drug: Bone marrow mesenchymal stem cells (low dose)
- Phase 1: Medium Dose Group (Experimental): The trial group with a low dose (2.0×10^6 cells/kg) will first enroll one subject, who will be infused with single dose CG-BM1 and then observed for at least 28 days. The clinical data of the first subject will be reviewed by the SRC.
  * If the first subject in the low-dose trial group experiences DLT, enrollment will be suspended. After discussion, recommendations will be made. If the trial is to continue, two additional subjects will be enrolled for observation. If no DLT occurs, the dose trial group will need to enroll three more subjects.
  * If the first subject in the dose trial group does not experience DLT after 28 days, - the remaining two subjects in that dose trial group will be enrolled.
  Once all subjects in the dose trial group have completed the infusion and have been observed for 28 days, the clinical data of all subjects will be submitted to the SRC. After a comprehensive evaluation, the SRC will provide recommendations for dose escalation.
  Interventions: Drug: Bone marrow mesenchymal stem cells (medium dose)
- Phase 1: High Dose Group (Experimental): The trial group with a low dose (4.0×10^6 cells/kg) will first enroll one subject, who will be infused with single dose CG-BM1 and then observed for at least 28 days. The clinical data of the first subject will be reviewed by the SRC.
  * If the first subject in the low-dose trial group experiences DLT, enrollment will be suspended. After discussion, recommendations will be made. If the trial is to continue, two additional subjects will be enrolled for observation. If no DLT occurs, the dose trial group will need to enroll three more subjects.
  * If the first subject in the dose trial group does not experience DLT after 28 days, - the remaining two subjects in that dose trial group will be enrolled.
  Once all subjects in the dose trial group have completed the infusion and have been observed for 28 days, the clinical data of all subjects will be submitted to the SRC. After a comprehensive evaluation, the SRC will provide recommendations for dose escalation.
  Interventions: Drug: Bone marrow mesenchymal stem cells (high dose)

INTERVENTIONS:
Drug: Bone marrow mesenchymal stem cells (low dose) — Administered intravenously. For phase I: single infusion, 1.0×10^6 cells/kg. For phase II: 1.0×10^6 cells /kg once a week for a total of 4 times.
  Other Names: CG-BM1
  Arms: Phase 1: Low Dose Group; Phase 2: Low Dose Group
Drug: Solvent of CG-BM1 — Administered intravenously, once a week for a total of 4 doses.
  Arms: Phase 2: Placebo Control
Drug: Bone marrow mesenchymal stem cells (medium dose) — Administered intravenously. For phase I: single infusion, 2.0×10^6 cells /kg. For phase II: 2.0×10^6 cells /kg once a week for a total of 4 times.
  Arms: Phase 1: Medium Dose Group; Phase 2: Medium Dose Group
Drug: Bone marrow mesenchymal stem cells (high dose) — Administered intravenously. For phase I: single infusion, 4×10^6 cells /kg.
  Arms: Phase 1: High Dose Group

SUMMARY:
The goal of this clinical trial is to learn if CG-BM1 Allogeneic Human Bone Marrow Mesenchymal Stem Cell Injection (hereinafter referred to as CG-BM1) can treat acute-on-chronic liver failure (ACLF) patients. Main purposes of this clinical trial are:

* To evaluate the safety and tolerability of CG-BM1 for the treatment of adult patients with ACLF.
* To observe the preliminary effectiveness of CG-BM1 in treating adult ACLF patients, and to provide a basis for subsequent clinical trial protocol design.

DETAILED DESCRIPTION:
CG-BM1 is a bone marrow mesenchymal stem cell product independently developed by Guangzhou Cellgenes Biotechnology Co., Ltd. The active ingredient of CG-BM1 is human bone marrow mesenchymal stem cell, which is derived from bone marrow donated by healthy adults and prepared into stem cell injection under aseptic conditions. CG-BM1 is the first bone marrow mesenchymal stem cell (BMSC) therapeutic drug for the treatment of ACLF in China. Preclinical data showed that CG-BM1 has the ability to immunomodulate, inhibit the secretion of pro-inflammatory factors by immune cells, and up-regulate the level of anti-inflammatory factors, which can significantly improve the liver function, reduce the inflammatory response, and reverse hepatic fibrosis in ACLF animal models, and the results of the study suggest that it is safe and effective, supporting its further clinical development. The purpose of this study was to evaluate the safety and tolerability of CG-BM1 for the treatment of patients with ACLF, as well as to evaluate the preliminary efficacy of CG-BM1 for the treatment of patients with ACLF.

The study was divided into 2 phases, the first with an open-labeled, dose-escalation design; the second with a multicenter, randomized, double-blind, placebo-controlled design. Phase I: Patients was divided into three dose groups using a traditional "3+3" design. 3-6 subjects were enrolled in each dose. Phase II: Multiple-dose, randomized, double-blind, placebo-controlled trial. Based on the results of the phase I trial, two dose groups were selected for phase II.

A total of 90 subjects were enrolled and randomized 1:1:1. The experiment group received CG-BM1 + conventional treatment regimen, and the control group received placebo + conventional treatment regimen.

ELIGIBILITY:
Phase I:

Inclusion Criteria:

1. Voluntarily participate in the clinical study. The patient or legal guardian fully understands and is informed about the study and signs an informed consent form. Willing to follow and be able to complete all trial procedures.
2. Age ≥18 years old, male or female.
3. Diagnostic criteria in accordance with the Guidelines for Diagnosis and Treatment of Liver Failure (2018 edition) issued by the Liver Failure and Artificial Liver Group of the Infectious Diseases Branch of the Chinese Medical Association and the Liver Disease Branch of the Chinese Medical Association Diagnostic criteria, specific indicators include 1) Suffering from the basis of chronic liver disease; 2) Serum TBIL 171 μ mol/l or mean daily rise ≥17.1 μmol/L; 3) Meeting any of the following three: i. Having a bleeding tendency; ii. Comorbid hepatic encephalopathy; iii. Comorbid hepatorenal syndrome.
4. The cause of liver failure is unlimited.
5. Model for End Stage Liver Disease (MELD) score under 30.
6. No conception (or conception of sexual partner) during the study period (from signing of informed consent to the last visit) and within 6 months after the last cell infusion; and childbearing, or breastfeeding potential, including:

   * Female subject with persistent spontaneous menopause >12 months or who have undergone sterilization (e.g., tubal ligation or bilateral oophorectomy or hysterectomy).
   * Non-menopausal female subject with a negative serum pregnancy test within 7 days prior to the first cellular infusion. Sign an informed consent and willingness to use one of the following effective methods of contraception, including intrauterine device (IUD), tubal ligation, double barrier method (condom, vaginal diaphragm, spermicide) and spermicide for the male partner, but does not include oral contraceptives, for a period of 6 months after the last cellular infusion.
   * Male subjects who are willing to use one or more effective methods of contraception, including vasectomy, double-barrier methods, use of the pill by the female partner, intrauterine devices or tubal ligation from the time of the first infusion until 6 months after the last infusion.
   * Male or non-menopausal female subjects who do not have, or are willing to not have sexual intercourse during the study and for 6 months after the last cell infusion.

Exclusion Criteria:

1. Be allergic to known components of the drug (the main component of the product is bone marrow mesenchymal stem cells, excipients include dimethyl sulfoxide, human albumin) or other history of severe allergy.
2. Patients with severe infections such as septic shock.
3. Patients with gastrointestinal bleeding at the time of screening.
4. Hepatic encephalopathy grade 4.
5. Concurrent failure of 3 or more organs (liver failure defined as TBiL ≥12 mg/dl, renal failure defined as creatinine ≥2.0 mg/dl, coagulation failure defined as INR ≥2.5, cerebral failure defined as hepatic encephalopathy grades 3-4, circulatory failure defined by use of vasoactive drugs, and respiratory failure was defined as PaO2 /FiO2 ≤200 or SpO2 /FiO2 ≤214 or mechanical ventilation)
6. Pregnancy or breastfeeding.
7. Previous history of malignant tumors.
8. Imaging suggestive of intrahepatic nodular space-occupying lesions.
9. A history of immunodeficiency, including HIV-positive, or other acquired or congenital immunodeficiency diseases.
10. Patients with previous liver transplantation.
11. Deep vein thrombosis at screening or history of pulmonary embolism within 3 months prior to screening.
12. Patients with pulmonary hypertension.
13. History of myocardial infarction within 6 months.
14. Previous stem cell therapy.
15. Participation in another interventional clinical trial within 3 months or 5 half-lives (for experimental drug interventions only, whichever is longer) prior to infusion.
16. Any other factors that, in the judgment of the investigator, make the subject inappropriate for participation in this trial.

Phase II:

Inclusion Criteria:

Inclusion Criteria:

1. Voluntarily participate in the clinical study. The patient or legal guardian fully understands and is informed about the study and signs an informed consent form. Willing to follow and be able to complete all trial procedures.
2. Age ≥18 years old, male or female.
3. Diagnostic criteria in accordance with the Guidelines for Diagnosis and Treatment of Liver Failure (2018 edition) issued by the Liver Failure and Artificial Liver Group of the Infectious Diseases Branch of the Chinese Medical Association and the Liver Disease Branch of the Chinese Medical Association Diagnostic criteria, specific indicators include 1) Suffering from the basis of chronic liver disease; 2) Serum TBIL 171 μ mol/l or mean daily rise ≥17.1 μmol/L; 3) Meeting any of the following three: i. Having a bleeding tendency; ii. Comorbid hepatic encephalopathy; iii. Comorbid hepatorenal syndrome.
4. The cause of liver failure is Hepatitis B.
5. Model for End Stage Liver Disease (MELD) score under 30.
6. No conception (or conception of sexual partner) during the study period (from signing of informed consent to the last visit) and within 6 months after the last cell infusion; and childbearing, or breastfeeding potential, including:

   * Female subject with persistent spontaneous menopause >12 months or who have undergone sterilization (e.g., tubal ligation or bilateral oophorectomy or hysterectomy).
   * Non-menopausal female subject with a negative serum pregnancy test within 7 days prior to the first cellular infusion. Sign an informed consent and willingness to use one of the following effective methods of contraception, including intrauterine device (IUD), tubal ligation, double barrier method (condom, vaginal diaphragm, spermicide) and spermicide for the male partner, but does not include oral contraceptives, for a period of 6 months after the last cellular infusion.
   * Male subjects who are willing to use one or more effective methods of contraception, including vasectomy, double-barrier methods, use of the pill by the female partner, intrauterine devices or tubal ligation from the time of the first infusion until 6 months after the last infusion.
   * Male or non-menopausal female subjects who do not have, or are willing to not have sexual intercourse during the study and for 6 months after the last cell infusion.

Exclusion Criteria:

1. Be allergic to known components of the drug (the main component of the product is bone marrow mesenchymal stem cells, excipients include dimethyl sulfoxide, human albumin) or other history of severe allergy.
2. Patients with severe infections such as septic shock.
3. Patients with gastrointestinal bleeding at the time of screening.
4. Hepatic encephalopathy grade 4.
5. Concurrent failure of 3 or more organs (liver failure defined as TBiL ≥12 mg/dl, renal failure defined as creatinine ≥2.0 mg/dl, coagulation failure defined as INR ≥2.5, cerebral failure defined as hepatic encephalopathy grades 3-4, circulatory failure defined by use of vasoactive drugs, and respiratory failure was defined as PaO2 /FiO2 ≤200 or SpO2 /FiO2 ≤214 or mechanical ventilation)
6. Pregnancy or breastfeeding.
7. Previous history of malignant tumors.
8. Imaging suggestive of intrahepatic solid nodal space-occupying lesions and which the investigator determines may compromise subject safety.
9. Received artificial liver therapy within 7 days prior to first dose.
10. A history of immunodeficiency, including HIV-positive, or other acquired or congenital immunodeficiency diseases.
11. Patients with previous liver transplantation.
12. Deep vein thrombosis at screening or history of pulmonary embolism within 3 months prior to screening.
13. Patients with pulmonary hypertension.
14. History of myocardial infarction within 6 months.
15. Previous stem cell therapy.
16. Participation in another interventional clinical trial within 3 months or 5 half-lives (for experimental drug interventions only, whichever is longer) prior to infusion.
17. Any other factors that, in the judgment of the investigator, make the subject inappropriate for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence of CG-BM1-related dose-limiting toxicity (DLT) events | From first dose to 180 days after the first dose.
  Incidence of CG-BM1-related DLT events.
Phase I: Adverse event related to CG-BM1 treatment | From first dose to 180 days after the first dose.
  Any adverse event related to CG-BM1 treatment that occurred during the study period.
Phase II: Liver transplant-free survival | 90 day after the first dose.
  90-day liver transplant-free survival.

SECONDARY OUTCOMES:
Phase I: Liver transplant-free survival | 28 day, 90 day, and 180 days after the first dose.
  28-day, 90-day, and 180-day liver transplant-free survival.
Phase I: Changes of aspartate aminotransferase (AST) | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days, 90 days after the first dose.
  Amount of increase or decrease in serum AST.
Phase I: Changes of alanine aminotransferase (ALT) | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days, 90 days after the first dose.
  Amount of increase or decrease in serum ALT.
Phase I: Changes of albumin | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days, 90 days after the first dose.
  Amount of increase or decrease in serum albumin.
Phase I: Changes of alkaline phosphatase (ALP) | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days, 90 days after the first dose.
  Amount of increase or decrease in serum ALP.
Phase I: Changes of γ-glutamyl transpeptidase (GGT) | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days, 90 days after the first dose.
  Amount of increase or decrease in serum GGT.
Phase I: Changes of total bilirubin (TBil) | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days, 90 days after the first dose.
  Amount of increase or decrease in serum TBil.
Phase I: Changes of international normalized ratio (INR) | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days, 90 days after the first dose.
  Amount of increase or decrease in INR.
Phase I: Changes in liver stiffness measurement (LSM) values | Pre-treatment, 14 days, 28 days, 60 days, 90 days after the first dose.
  Changes in LSM values measured by transient elastography (TE).
Phase I: Changes of 15-minute retention rate obtained by indocyanine green (ICG) retention test | Pre-treatment, 7 days, 14 days, 28 days, 60 days, 90 days after the first dose.
  Changes of 15-minute retention rate obtained by indocyanine green (ICG) retention test. Inject indocyanine green (ICG) rapidly into a peripheral vein on one side of the patient at a dose of 0.5mg/kg body weight, and start timing immediately after the injection. After 15 minutes, draw 2ml of blood from the opposite side peripheral vein, separate the serum, and measure the concentration of indocyanine green using a spectrophotometer. Calculate the indocyanine green retention rate at 15 minutes using the following formula: ICG Retention Rate (%) = (C15 mg% ÷ 1 mg%) × 100%.
Phase I: Complication rate | 180 days after the first dose.
  Complication rate within 180 days.
Phase I: Changes in chronic liver failure consortium organ failure score (CLIF-C OFs) | Pre-treatment, 3 days, 7 days, 14 days, 28 days, 60 days, 90 days after the first dose.
  Changes in CLIF-C OFs. Each organ system is scored on a scale to generate the overall CLIF-C OF score, ranging from 0 to 18. The higher the CLIF C OF score, the poorer the prognosis for the patient, which means a higher short-term mortality rate.
Phase I: Changes in Model for end-stage liver disease (MELD) score | Pre-treatment, 3 days, 7 days, 14 days, 28 days, 60 days, 90 days after the first dose.
  MELDScore = 10 * ((0.957 * ln(Creatinine)) + (0.378 * ln(Bilirubin)) + (1.12 * ln(INR))) + 6.43. An increase in the MELD score indicates worse liver function, poorer prognosis, and a higher urgency for liver transplantation.
Phase I: Anti-human histocompatibility antigen antibody (HLA-Ab) positivity rate | Pre-treatment, 28 days, 60 days after the first dose.
  Serum HLA-Ab positivity rate.
Phase I: Serum Interleukin-6 (IL-6) levels | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days after the first dose.
  Serum IL-6 levels.
Phase I: Serum tumor necrosis factor-α (TNF-α) levels | Pre-treatment, 3 days, 7 days, 14 days, 21 days, 28 days after the first dose.
  Serum TNF-α levels.
Phase II: Adverse event related to CG-BM1 treatment | From first dose to 180 days after the first dose.
  Any adverse event related to CG-BM1 treatment that occurred during the study period.
Phase II: Liver transplant-free survival | 28 days, 180 days after the first dose.
  28-day, 180-day liver transplant-free survival.
Phase II: Changes in Model for end-stage liver disease (MELD) score | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  MELDScore = 10 * ((0.957 * ln(Creatinine)) + (0.378 * ln(Bilirubin)) + (1.12 * ln(INR))) + 6.43. An increase in the MELD score indicates worse liver function, poorer prognosis, and a higher urgency for liver transplantation.
Phase II: Changes in chronic liver failure consortium organ failure score (CLIF-C OFs) | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Changes in CLIF-C OFs. Each organ system is scored on a scale to generate the overall CLIF-C OF score, ranging from 0 to 18. The higher the CLIF-C OF score, the poorer the prognosis for the patient, which means a higher short-term mortality rate.
Phase II: Complication rate | 180 days after the first dose.
  Complication rate within 180 days. Including: cerebral edema, hepatic encephalopathy, infection, hyponatremia, refractory ascites, acute kidney injury, hepatorenal syndrome, hemorrhage, hepatopulmonary syndrome.
Phase II: Changes of aspartate aminotransferase (AST) | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Amount of increase or decrease in serum AST.
Phase II: Changes of alanine aminotransferase (ALT) | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Amount of increase or decrease in serum ALT.
Phase II: Changes of albumin | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Amount of increase or decrease in serum albumin.
Phase II: Changes of alkaline phosphatase (ALP) | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Amount of increase or decrease in serum ALP.
Phase II: Changes of γ-glutamyl transpeptidase (GGT) | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Amount of increase or decrease in serum GGT.
Phase II: Changes of total bilirubin (TBil) | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Amount of increase or decrease in serum TBil.
Phase II: Changes of international normalized ratio (INR) | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Amount of increase or decrease in INR.
Phase II: Changes in liver stiffness measurement (LSM) values | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Changes in LSM values measured by transient elastography (TE).
Phase II: Changes of 15-minute retention rate obtained by indocyanine green (ICG) retention test | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Changes of 15-minute retention rate obtained by indocyanine green (ICG) retention test. Inject indocyanine green (ICG) rapidly into a peripheral vein on one side of the patient at a dose of 0.5mg/kg body weight, and start timing immediately after the injection. After 15 minutes, draw 2ml of blood from the opposite side peripheral vein, separate the serum, and measure the concentration of indocyanine green using a spectrophotometer. Calculate the indocyanine green retention rate at 15 minutes using the following formula: ICG Retention Rate (%) = (C15 mg% ÷ 1 mg%) × 100%.
Phase II: Anti-human histocompatibility antigen antibody (HLA-Ab) positivity rate | Pre-treatment, 28 days, 90 days after the first dose.
  Serum HLA-Ab positivity rate.
Phase II: Serum Interleukin-6 (IL-6) levels | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Serum IL-6 levels.
Phase II: Serum tumor necrosis factor-α (TNF-α) levels | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Serum TNF-α levels.
Phase II: Serum hepatocyte growth factor (HGF) levels | Pre-treatment, 28 days, 60 days, 90 days, 180 days after the first dose.
  Serum HGF levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klopp AH, Gupta A, Spaeth E, Andreeff M, Marini F 3rd. Concise review: Dissecting a discrepancy in the literature: do mesenchymal stem cells support or suppress tumor growth? Stem Cells. 2011 Jan;29(1):11-9. doi: 10.1002/stem.559. PMID 21280155
- [Background] Kaipe H, Carlson LM, Erkers T, Nava S, Mollden P, Gustafsson B, Qian H, Li X, Hashimoto T, Sadeghi B, Alheim M, Ringden O. Immunogenicity of decidual stromal cells in an epidermolysis bullosa patient and in allogeneic hematopoietic stem cell transplantation patients. Stem Cells Dev. 2015 Jun 15;24(12):1471-82. doi: 10.1089/scd.2014.0568. Epub 2015 Mar 13. PMID 25658253
- [Background] Hare JM, Fishman JE, Gerstenblith G, DiFede Velazquez DL, Zambrano JP, Suncion VY, Tracy M, Ghersin E, Johnston PV, Brinker JA, Breton E, Davis-Sproul J, Schulman IH, Byrnes J, Mendizabal AM, Lowery MH, Rouy D, Altman P, Wong Po Foo C, Ruiz P, Amador A, Da Silva J, McNiece IK, Heldman AW, George R, Lardo A. Comparison of allogeneic vs autologous bone marrow-derived mesenchymal stem cells delivered by transendocardial injection in patients with ischemic cardiomyopathy: the POSEIDON randomized trial. JAMA. 2012 Dec 12;308(22):2369-79. doi: 10.1001/jama.2012.25321. PMID 23117550
- [Background] Poncelet AJ, Vercruysse J, Saliez A, Gianello P. Although pig allogeneic mesenchymal stem cells are not immunogenic in vitro, intracardiac injection elicits an immune response in vivo. Transplantation. 2007 Mar 27;83(6):783-90. doi: 10.1097/01.tp.0000258649.23081.a3. PMID 17414713
- [Background] Ra JC, Shin IS, Kim SH, Kang SK, Kang BC, Lee HY, Kim YJ, Jo JY, Yoon EJ, Choi HJ, Kwon E. Safety of intravenous infusion of human adipose tissue-derived mesenchymal stem cells in animals and humans. Stem Cells Dev. 2011 Aug;20(8):1297-308. doi: 10.1089/scd.2010.0466. Epub 2011 Mar 17. PMID 21303266
- [Background] Zhang K, Sun H, Cao H, Jia Y, Shu X, Cao H, Zhang Y, Yang X. The impact of recipient age on the effects of umbilical cord mesenchymal stem cells on HBV-related acute-on-chronic liver failure and liver cirrhosis. Stem Cell Res Ther. 2021 Aug 20;12(1):466. doi: 10.1186/s13287-021-02544-x. PMID 34416908
- [Background] Xu WX, He HL, Pan SW, Chen YL, Zhang ML, Zhu S, Gao ZL, Peng L, Li JG. Combination Treatments of Plasma Exchange and Umbilical Cord-Derived Mesenchymal Stem Cell Transplantation for Patients with Hepatitis B Virus-Related Acute-on-Chronic Liver Failure: A Clinical Trial in China. Stem Cells Int. 2019 Feb 4;2019:4130757. doi: 10.1155/2019/4130757. eCollection 2019. PMID 30863450
- [Background] Li YH, Xu Y, Wu HM, Yang J, Yang LH, Yue-Meng W. Umbilical Cord-Derived Mesenchymal Stem Cell Transplantation in Hepatitis B Virus Related Acute-on-Chronic Liver Failure Treated with Plasma Exchange and Entecavir: a 24-Month Prospective Study. Stem Cell Rev Rep. 2016 Dec;12(6):645-653. doi: 10.1007/s12015-016-9683-3. PMID 27687792
- [Background] Shi M, Zhang Z, Xu R, Lin H, Fu J, Zou Z, Zhang A, Shi J, Chen L, Lv S, He W, Geng H, Jin L, Liu Z, Wang FS. Human mesenchymal stem cell transfusion is safe and improves liver function in acute-on-chronic liver failure patients. Stem Cells Transl Med. 2012 Oct;1(10):725-31. doi: 10.5966/sctm.2012-0034. Epub 2012 Oct 11. PMID 23197664
- [Background] Schacher FC, Martins Pezzi da Silva A, Silla LMDR, Alvares-da-Silva MR. Bone Marrow Mesenchymal Stem Cells in Acute-on-Chronic Liver Failure Grades 2 and 3: A Phase I-II Randomized Clinical Trial. Can J Gastroenterol Hepatol. 2021 Aug 4;2021:3662776. doi: 10.1155/2021/3662776. eCollection 2021. PMID 34395335
- [Background] Peng L, Xie DY, Lin BL, Liu J, Zhu HP, Xie C, Zheng YB, Gao ZL. Autologous bone marrow mesenchymal stem cell transplantation in liver failure patients caused by hepatitis B: short-term and long-term outcomes. Hepatology. 2011 Sep 2;54(3):820-8. doi: 10.1002/hep.24434. Epub 2011 Jul 14. PMID 21608000
- [Background] Lin BL, Chen JF, Qiu WH, Wang KW, Xie DY, Chen XY, Liu QL, Peng L, Li JG, Mei YY, Weng WZ, Peng YW, Cao HJ, Xie JQ, Xie SB, Xiang AP, Gao ZL. Allogeneic bone marrow-derived mesenchymal stromal cells for hepatitis B virus-related acute-on-chronic liver failure: A randomized controlled trial. Hepatology. 2017 Jul;66(1):209-219. doi: 10.1002/hep.29189. Epub 2017 May 27. PMID 28370357
- [Background] Zheng J, Chen L, Lu T, Zhang Y, Sui X, Li Y, Huang X, He L, Cai J, Zhou C, Liang J, Chen G, Yao J, Yang Y. MSCs ameliorate hepatocellular apoptosis mediated by PINK1-dependent mitophagy in liver ischemia/reperfusion injury through AMPKalpha activation. Cell Death Dis. 2020 Apr 20;11(4):256. doi: 10.1038/s41419-020-2424-1. PMID 32312955
- [Background] Zhao S, Liu Y, Pu Z. Bone marrow mesenchymal stem cell-derived exosomes attenuate D-GaIN/LPS-induced hepatocyte apoptosis by activating autophagy in vitro. Drug Des Devel Ther. 2019 Aug 19;13:2887-2897. doi: 10.2147/DDDT.S220190. eCollection 2019. PMID 31695322
- [Background] Naji A, Eitoku M, Favier B, Deschaseaux F, Rouas-Freiss N, Suganuma N. Biological functions of mesenchymal stem cells and clinical implications. Cell Mol Life Sci. 2019 Sep;76(17):3323-3348. doi: 10.1007/s00018-019-03125-1. Epub 2019 May 4. PMID 31055643
- [Background] Le Blanc K, Tammik C, Rosendahl K, Zetterberg E, Ringden O. HLA expression and immunologic properties of differentiated and undifferentiated mesenchymal stem cells. Exp Hematol. 2003 Oct;31(10):890-6. doi: 10.1016/s0301-472x(03)00110-3. PMID 14550804
- [Background] Horwitz EM, Le Blanc K, Dominici M, Mueller I, Slaper-Cortenbach I, Marini FC, Deans RJ, Krause DS, Keating A; International Society for Cellular Therapy. Clarification of the nomenclature for MSC: The International Society for Cellular Therapy position statement. Cytotherapy. 2005;7(5):393-5. doi: 10.1080/14653240500319234. PMID 16236628
- [Background] Li J, Liang X, Jiang J, Yang L, Xin J, Shi D, Lu Y, Li J, Ren K, Hassan HM, Zhang J, Chen P, Yao H, Li J, Wu T, Jin L, Ye P, Li T, Zhang H, Sun S, Guo B, Zhou X, Cai Q, Chen J, Xu X, Huang J, Hao S, He J, Xin S, Wang D, Trebicka J, Chen X, Li J; Chinese Group on the Study of Severe Hepatitis B (COSSH). PBMC transcriptomics identifies immune-metabolism disorder during the development of HBV-ACLF. Gut. 2022 Jan;71(1):163-175. doi: 10.1136/gutjnl-2020-323395. Epub 2021 Jan 11. PMID 33431576
- [Background] Wu T, Li J, Shao L, Xin J, Jiang L, Zhou Q, Shi D, Jiang J, Sun S, Jin L, Ye P, Yang L, Lu Y, Li T, Huang J, Xu X, Chen J, Hao S, Chen Y, Xin S, Gao Z, Duan Z, Han T, Wang Y, Gan J, Feng T, Pan C, Chen Y, Li H, Huang Y, Xie Q, Lin S, Li L, Li J; Chinese Group on the Study of Severe Hepatitis B (COSSH).. Development of diagnostic criteria and a prognostic score for hepatitis B virus-related acute-on-chronic liver failure. Gut. 2018 Dec;67(12):2181-2191. doi: 10.1136/gutjnl-2017-314641. Epub 2017 Sep 19. PMID 28928275
- [Background] Shi Y, Yang Y, Hu Y, Wu W, Yang Q, Zheng M, Zhang S, Xu Z, Wu Y, Yan H, Chen Z. Acute-on-chronic liver failure precipitated by hepatic injury is distinct from that precipitated by extrahepatic insults. Hepatology. 2015 Jul;62(1):232-42. doi: 10.1002/hep.27795. Epub 2015 Apr 25. PMID 25800029
- [Background] Lin B, Pan CQ, Xie D, Xie J, Xie S, Zhang X, Wu B, Lin C, Gao Z. Entecavir improves the outcome of acute-on-chronic liver failure due to the acute exacerbation of chronic hepatitis B. Hepatol Int. 2013 Jun;7(2):460-7. doi: 10.1007/s12072-012-9415-y. Epub 2013 Feb 11. PMID 26201778
- [Background] Mezzano G, Juanola A, Cardenas A, Mezey E, Hamilton JP, Pose E, Graupera I, Gines P, Sola E, Hernaez R. Global burden of disease: acute-on-chronic liver failure, a systematic review and meta-analysis. Gut. 2022 Jan;71(1):148-155. doi: 10.1136/gutjnl-2020-322161. Epub 2021 Jan 12. PMID 33436495
- [Background] Sarin SK, Choudhury A, Sharma MK, Maiwall R, Al Mahtab M, Rahman S, Saigal S, Saraf N, Soin AS, Devarbhavi H, Kim DJ, Dhiman RK, Duseja A, Taneja S, Eapen CE, Goel A, Ning Q, Chen T, Ma K, Duan Z, Yu C, Treeprasertsuk S, Hamid SS, Butt AS, Jafri W, Shukla A, Saraswat V, Tan SS, Sood A, Midha V, Goyal O, Ghazinyan H, Arora A, Hu J, Sahu M, Rao PN, Lee GH, Lim SG, Lesmana LA, Lesmana CR, Shah S, Prasad VGM, Payawal DA, Abbas Z, Dokmeci AK, Sollano JD, Carpio G, Shresta A, Lau GK, Fazal Karim M, Shiha G, Gani R, Kalista KF, Yuen MF, Alam S, Khanna R, Sood V, Lal BB, Pamecha V, Jindal A, Rajan V, Arora V, Yokosuka O, Niriella MA, Li H, Qi X, Tanaka A, Mochida S, Chaudhuri DR, Gane E, Win KM, Chen WT, Rela M, Kapoor D, Rastogi A, Kale P, Rastogi A, Sharma CB, Bajpai M, Singh V, Premkumar M, Maharashi S, Olithselvan A, Philips CA, Srivastava A, Yachha SK, Wani ZA, Thapa BR, Saraya A, Shalimar, Kumar A, Wadhawan M, Gupta S, Madan K, Sakhuja P, Vij V, Sharma BC, Garg H, Garg V, Kalal C, Anand L, Vyas T, Mathur RP, Kumar G, Jain P, Pasupuleti SSR, Chawla YK, Chowdhury A, Alam S, Song DS, Yang JM, Yoon EL; APASL ACLF Research Consortium (AARC) for APASL ACLF working Party.. Acute-on-chronic liver failure: consensus recommendations of the Asian Pacific association for the study of the liver (APASL): an update. Hepatol Int. 2019 Jul;13(4):353-390. doi: 10.1007/s12072-019-09946-3. Epub 2019 Jun 6. PMID 31172417